CLINICAL TRIAL: NCT06254339
Title: The Effect of MBS on Outcomes and Reduction of the 10-year and Lifetime Risks of MACE: Analysis of 224 Patients Undergoing OAGB and DJB-SG During a 7-year Period.
Brief Title: Effects of OAGB and DJB-SG on 10-year and Lifetime Risks of MACE
Status: Completed | Type: Observational
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Kuo-Feng Hsu, Principal investigator, National Defense Medical Center, Taiwan
Other Study IDs: B202105089
Record Dates: First submitted 2024-01-24; First posted 2024-02-12 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Obesity
Keywords: One-anastomosis gastric bypass; Duodenal-jejunal bypass with sleeve gastrectomy; Major adverse cardiovascular events; Type 2 diabetes mellitus; Obesity; Comorbidities
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OAGB cohort: Application of One-anastomosis gastric bypass (OAGB) procedure stated in IFSO/ASMBS.
  Interventions: Procedure: OAGB
- DJB-SG cohort: Application of Duodenojejunal bypass with sleeve gastrectomy (DJB-SG)) procedure stated in IFSO/ASMBS.
  Interventions: Procedure: DJB-SG

INTERVENTIONS:
Procedure: OAGB — using OAGB procedure as metabolic bariatric surgery
  Groups: OAGB cohort
Procedure: DJB-SG — using DJB-SG procedure as metabolic bariatric surgery
  Groups: DJB-SG cohort

SUMMARY:
Metabolic bariatric surgery (MBS) has demonstrated its efficacy in achieving sustainable weight loss and alleviating associated comorbidities. The primary objective of our investigation is to assess the long-term impact and sustainability of weight loss, the remission of T2D as well as risk prediction of cardiovascular events following MBS concerning one-anastomosis gastric bypass (OAGB) and duodenojejunal bypass with sleeve gastrectomy (DJB-SG).

DETAILED DESCRIPTION:
Metabolic bariatric surgery (MBS) offers enduring weight reduction and alleviation of obesity-related comorbidities, including dyslipidemia, type 2 diabetes (T2D), hypertension (HTN), and major adverse cardiovascular events (MACE). Long-term data on one anastomosis gastric bypass (OAGB) and duodenal-jejunal bypass with sleeve gastrectomy (DJB-SG) is lacking, necessitating this investigation. In this multicenter prospectively-collected retrospective observational study, patients with complete follow-up data at various intervals up to 3 years after surgery were included in the final analysis. The study's primary focus was to evaluate the long-term safety, efficacy, and durability of OAGB and DJB-SG in promoting weight loss and T2D remission. Additionally, changes in 10-year and lifetime risks of MACE before and 3-year after surgery were assessed using the Taiwan MACE risk prediction model and the China-PAR project model based on Taiwan national electronic health records and a large Chinese participant dataset, respectively.

Hypothesis: This study contributes to providing valuable information in terms of the impacts of OAGB and DJB-SG on patients with obesity and associated diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose BMI≧37.5 kg/m2 or patients whose BMI≧32.5 kg/m2 and have concurrent high-risk comorbidities, such as hypertension, obstructive sleep apnea, HbA1c≧7.5% after anti-diabetic medication treatment, etc;
* The patients have been treated with lifestyle intervention, including increase in physical activity and change in diet, for more than 6 months;
* Age between 20 and 65 years old;
* Patients without other endocrinological causes that result in morbid obesity;
* Patients without substance use, alcohol use and other psychiatric disorders;
* The integrity of the patient's mental status is approved by the psychiatrist.

Exclusion Criteria:

* Patients who did not complete 3-year follow-up
* Patients who are not eligible for surgery

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Taiwanese adult patients, whose age are between 20 and 65 years old, with obesity and/or cormobidities and metabolic disorders, such as type 2 diabetes mellitus, hypertension, dyslipidemia, obstructive sleep apnea, etc.
Sampling Method: Non-Probability Sample
Enrollment: 830 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 3 years
  Weight reduction
Diabetes | 3 years
  HbA1c change
Hypertension | 3 years
  Blood pressure (SBP/BP change)
Dyslipidemia | 3 years
  TG, T-CHO, LDL, HDL change

SECONDARY OUTCOMES:
Taiwan MACE risk prediction model | 10 years
  A 10-year MACE risk prediction model developed with Taiwan national data and death registry.
The China-PAR project model | 10 years
  A 10-year and lifetime prediction model for atherosclerotic cardiovascular disease risk in Chinese population, developed within the context of the Chinese population on a national scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mu-Xian Yu, MD, Study Chair — Tri-Service General Hospital, NDMC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bluher M. Obesity: global epidemiology and pathogenesis. Nat Rev Endocrinol. 2019 May;15(5):288-298. doi: 10.1038/s41574-019-0176-8. PMID 30814686
- [Background] Powell-Wiley TM, Poirier P, Burke LE, Despres JP, Gordon-Larsen P, Lavie CJ, Lear SA, Ndumele CE, Neeland IJ, Sanders P, St-Onge MP; American Heart Association Council on Lifestyle and Cardiometabolic Health; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Epidemiology and Prevention; and Stroke Council. Obesity and Cardiovascular Disease: A Scientific Statement From the American Heart Association. Circulation. 2021 May 25;143(21):e984-e1010. doi: 10.1161/CIR.0000000000000973. Epub 2021 Apr 22. PMID 33882682
- [Background] Michaels AD, Mehaffey JH, Hawkins RB, Kern JA, Schirmer BD, Hallowell PT. Bariatric surgery reduces long-term rates of cardiac events and need for coronary revascularization: a propensity-matched analysis. Surg Endosc. 2020 Jun;34(6):2638-2643. doi: 10.1007/s00464-019-07036-x. Epub 2019 Aug 2. PMID 31376005